CLINICAL TRIAL: NCT03368261
Title: Epidemiology and Pathophysiological Mechanisms of Pulmonary Arterial Hypertension in SS and SC Children in Martinique and Guadeloupe.Three Years Follow up of a Cohort of Children Aged From 8 to 16 Years Old
Brief Title: Epidemiology and Pathophysiological Mechanisms of HTAP in SS and SC Children in Martinique and Guadeloupe.
Acronym: SAPOTILLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RBM-PAP-2009/69
Record Dates: First submitted 2017-12-01; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Sickle Cell Disease
Keywords: Pulmonary arterial hypertension; SCD; Epidemiology
MeSH Terms: conditions — Anemia, Sickle Cell; Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HTAP/ clinical complications in the sickle cell disease (Other): Supply epidemiological data on this detected HTAP, and allow the characterization of the clinico-biological paintings and the mortality which are associated to them.
  Interventions: Other: HTAP/ clinical complications in the sickle cell disease

INTERVENTIONS:
Other: HTAP/ clinical complications in the sickle cell disease — At the inclusion in our study the diagnosis of PAH will be performed by transthoracic Doppler-echocardiograms in a group of 306 children (aged between 8 to 16 years old) with either SS or SC genotype with similar medical caring, to avoid a known selection bias. These patients will be followed during a 3 years longitudinal period. The occurrence of the clinical specific complications associated with SCD (acute chest syndrome, painful vaso occlusive crisis, septicemia and stroke) and the observed mortality rate of our children group, will be compared in patients groups stratified according to the occurrence of PAH. The expression of several molecular and cellular genetic biomarkers potentially associated with this complication will also be studied.

SUMMARY:
pulmonary arterial hypertension (PAH) has been reported with a prevalence of approximately 30% in adult sickle cell disease (SCD) patients, with an increased mortality in SCD patients with PAH, compared with those without PAH. The identification of several hemolysis biomarkers such as lactate dehydrogenase, bilirubin, reticulocytes or hemoglobin level, has clearly documented a link between hemolysis and PAH. However, other physiopathological mechanisms may be involved to explain PAH in these patients, such as pulmonary thromboembolism, pulmonary fibrosis or left heart diastolic and / or systolic dysfunction.

The investigators suggest studying HTAP in patient's presenting the most frequent both drepanocytic syndromes, SS and SC and homogeneous in their medical coverage and the association between HTAP risk and specific SCD complications.

DETAILED DESCRIPTION:
The primary aim of this study is to estimate the prevalence and the incidence of PAH in a population of SCD children (SS, SC) with similar medical caring, aged from 8 to 16 years old.

Unlike the important number of studies in SCD adults, very few SCD children studies were performed. None of these studies reported the mortality rate associated with PAH in children although the literature reported a decrease of this morbid-mortality comparing different medical caring of the patients. The investigators hypothesized that physiopathological mechanisms responsible for PAH had to be different in SCD children compared with adults, as most degenerative processes had no time enough to appear during children's lives. At the inclusion in our study the diagnosis of PAH will be performed by transthoracic Doppler-echocardiograms in a group of 306 children (aged between 8 to 16 years old) with either SS or SC genotype with similar medical caring, to avoid a known selection bias. These patients will be followed during a 3 years longitudinal period. The occurrence of the clinical specific complications associated with SCD (acute chest syndrome, painful vaso occlusive crisis, septicemia and stroke) and the observed mortality rate of our children group, will be compared in patients groups stratified according to the occurrence of PAH. The expression of several molecular and cellular genetic biomarkers potentially associated with this complication will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* children aged between 8 to 16 years old,
* SS homozygote or SC compound heterozygote, followed by the sickle cell centers of Guadeloupe and Martinique or by the pediatric department of the university hospital of Fort-de-France, identified by the systematic neonatal screening programs performed in Guadeloupe and Martinique or by other labeled centers, registered in the French medical social security national program, and for which the parental and the old children consent has been obtained.

Exclusion Criteria:

* other hemoglobinopathies, chronic transfusion therapy programs or treatments which affected the expression of the biomarkers studied (unless hydroxyurea treatment),
* recent blood transfusion or phlebotomies (less than 3 months);
* patients not at steady state,
* pregnancy or breast feeding,
* refusal of parental and old children consent.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 185 (Actual)
Dates: Start 2010-01-11 (Actual); Primary Completion 2013-10-02 (Actual); Study Completion 2016-10-17 (Actual)

PRIMARY OUTCOMES:
incidence of pulmonary arterial hypertension | Through study completion, an average of 5 years
  The primary outcome of the present study is to estimate the incidence of pulmonary arterial hypertension documented by the presence of tricuspid regurgitation jet velocity of at least 2.5 ms-1 by Doppler echocardiographic assessment.

SECONDARY OUTCOMES:
The association between PAH risk and specific SCD complications | Through study completion, an average of 5 years
  To determine the association between PAH risk and specific SCD complications (painful crisis, acute chest syndrome, severe infectious events, stroke, cerebral vasculopathy), expression of molecular (pro-PBN, nitrite/ nitrate compounds, sVCAM-1, sICAM-1, S- and P-selectine, plasmatic hemoglobin, ET-1, CD40L), cellular (microparticles, hemorheological parameters) biomarkers, and genetic markers (alpha-globin, type 3 NOS, endothélin-1, ACVRL1, BMPR2, BMP6).
  To determine if PAH is a risk factor of the clinical complications cited previously above and of mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Maryse ETIENNE-JULAN, Doctor specializing in SCD, Study Director — Hospital University Center of Pointe-à-Pitre
Locations (1):
- Hospital University Center of Martinique, Fort-de-France, Martinique